CLINICAL TRIAL: NCT07033351
Title: The Effect of Platelet Rich Fibrin Layers on Peri-implant Tissue Phenotype
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Mustansiriyah University (Other)
Responsible Party: Principal Investigator, Ahmed Mahir Tawfeeq Karakchi, Principal Investigator, Al-Mustansiriyah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUOSU-202131
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Dental Implant; Platelet Rich Fibrin; Keratinized Mucosa; Crestal Bone Loss
Keywords: Platelet-Rich Fibrin (PRF); Dental Implant; Keratinized Mucosa; Crestal Bone Level; Soft Tissue Healing
MeSH Terms: interventions — Prolactin-Releasing Hormone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcomes assessor was blinded to the group allocation to prevent bias during the evaluation of soft tissue width and crestal bone measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0 PRF (Active Comparator): Each implant placed in this group did NOT have PRF membrane placed over the implant.
  Interventions: Procedure: Dental implant placement without PRF
- 1 PRF (Experimental): Each implant placed in this group had ONE PRF membrane placed over the implant.
  Interventions: Biological: Single-layer PRF membrane application
- 3 PRF (Experimental): Each implant placed in this group had THTEE STACKED PRF membranes placed over the implant.
  Interventions: Biological: Triple-layer PRF membrane application

INTERVENTIONS:
Procedure: Dental implant placement without PRF — Standard dental implant placement procedure with flap elevation and suturing, without the application of any PRF membrane over the implant site.
  Arms: 0 PRF
Biological: Single-layer PRF membrane application — PRF membrane prepared via centrifugation is applied as a single layer over the implant site following implant placement before flap closure.
  Arms: 1 PRF
Biological: Triple-layer PRF membrane application — Three autologous PRF membranes prepared via centrifugation are stacked and applied as a 3-layer membrane over the implant site before flap closure.
  Arms: 3 PRF

SUMMARY:
The present investigation seeks to determine how varying quantities of Platelet-Rich Fibrin (PRF) membranes influence the repair of both gingival and osseous tissues adjacent to dental implants. A secondary objective is to establish whether the incorporation of PRF contributes to enhanced stability of the soft-tissue cover and more effective retention of alveolar bone over an extended period.

Central to the study are two specific inquiries: Does the application of PRF correlate with an increase in the width and thickness of keratinized mucosa surrounding the implant? Is there a dose-response relationship such that the use of multiple PRF layers yields superior maintenance of bone height compared with a single layer or no PRF at all?

To address these questions, clinicians will juxtapose three treatment groups: one receiving no PRF, another receiving a single membrane, and a third receiving a triple-layer graft. Healing parameters will be measured before surgery and again at 6-week and 12-week checkpoints, allowing direct appraisal of outcome changes across the comparative cohorts.

Each participant will ultimately be allotted to one of the experimental arms by random assignment, thus mitigating selection bias. Routine follow-up examinations and radiographic imaging, will be used to track healing progress.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or female) over 18 years of age.
* Partially edentulous spaces.
* No history of bone augmentation procedures in the implant site.
* Good oral health, as measured by:
* Calibrated gingival bleeding index (≤10%)
* O'Leary plaque index (<10%)

Exclusion Criteria:

* Bleeding disorders.
* Compromised immune systems.
* Excessive smoking or alcohol consumption.
* Poor oral hygiene.
* Diabetes.
* Inability to attend follow-up visits.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-06 (Actual); Study Completion 2025-06-06 (Actual)

PRIMARY OUTCOMES:
Ridge Width Changes (RW) | Baseline (preoperative), immediate postoperative, 6 weeks, and 12 weeks
  The changes in Ridge Width is measured at the reference points using a digital vernier caliper.
Bone Width (BW) | Baseline (preoperative), and 12 weeks postoperatively
  Measured in millimeters by subtracting the buccal and lingual mucosal thickness from the ridge width.
Change in width of keratinized tissue (KTW) | Baseline (preoperative), 6 weeks, and 12 weeks
  Measured in millimeters at the mid-buccal aspect of the implant site using an endodontic rotary file and digital vernier caliper.
Keratinized Tissue Thickness (KTT) | Baseline (preoperative), and 12 weeks postoperatively
  Measured in millimeters at the buccal, crestal and lingual reference points using a periodontal probe and a digital vernier caliper.
Radiographic Mucosal Thickness (RT) | Baseline (preoperative), immediate postoperative, 6 weeks, and 12 weeks
  Measured in millimeters on periapical radiographs using digital software from the crestal bone level to the crest of crestal oral mucosa 5 mm away from the height distal surface of the adjacent tooth on the mesial side of the implant.
Crestal Bone Height (BH) | Immediate postoperative, 6 weeks, and 12 weeks
  Measured in millimeters on periapical radiographs using digital software from the second serration on the mesial side of the implant to the crest of the bone.

SECONDARY OUTCOMES:
Plaque Index (PI) | Baseline (preoperative), 6 weeks, and 12 weeks
  O'Leary plaque index
Gingival Index (GI) | Baseline (preoperative), 6 weeks, and 12 weeks
  Gingival Bleeding Index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Mosul / College of Dentistry, Mosul, Nenavah, Iraq